CLINICAL TRIAL: NCT06659484
Title: Evaluation and Changes of Disability Mobility Risk Factors in Older Adults Aged 70 and Over and Integrated in "Well on My Legs" Prevention Program.
Brief Title: Health Data from Well on My Legs Program
Acronym: DS-BSSJ
Status: Active, not recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 1791
Record Dates: First submitted 2024-10-23; First posted 2024-10-26 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Sarcopenia; Frailty; Physical Inactivity; Fear; Falling
Keywords: Older Adults; Mobility disability; prevention program; exercise; nutrition
MeSH Terms: conditions — Sarcopenia; Frailty; Sedentary Behavior; Motor Activity | interventions — Physical Examination; Triiodothyronine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Evaluation of the concentration of various markers of undernutrition (albuminemia and pre-albuminemia), inflammation (CRP) and metabolism (calcium and vitamin D) at T0 (initial assessment) and T3 (after the exercise program at around 3 months)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Community-dwelling older adults assessed without mobility disability risk factors following initial: Community-dwelling older adults aged of >70y, screened at risk of mobility disability risk factors and assessed without any mobility disability risk factors. This group is not included for intervention and received lifestyle counselling to maintain habits. No follow-up is conducted in this group.
  Or community-dwelling older adults aged of >70y, screened with medical contraindication. This group is not included for intervention and oriented to other medical practitioners. No follow-up is conducted in this group.
  Interventions: Diagnostic Test: Assessment; Other: Multicomponent exercise program; Other: Follow-up at T3 + 6 months and T3 + 12 months
- Community-dwelling older adults assessed with mobility disability risk factors following initial ass: Community-dwelling older adults aged of >70y, screened at risk of mobility disability risk factors and assessed with at least 1 mobility disability risk factor. This group is included for 3 months exercise intervention. Follow-up is conducted at 3 months (T3) and from T3 at 6 months (phone call) and 12 months.
  Interventions: Diagnostic Test: Assessment

INTERVENTIONS:
Diagnostic Test: Assessment — Evaluation carried out during a day hospital at T0 (initial assessment) and T3 (after the exercise program at around 3 months) including:
  1. Clinical assessment by a geriatrician
     * Medical history; systematic search for symptomatic elements (asthenia, anorexia, weight loss); research into antecedents (chronic pathologies, etc.), treatments, lifestyle, eating habits, sedentary lifestyle,
     * Complete clinical examination: particularly of the musculoskeletal system, morphological data (weight and height, calf circumference), analysis of risk of falls,
     * Current medical treatments
     * Autonomy for basic activities (ADL), instrumental activities of daily living (IADL), visual disorders, hearing impairment, etc.
     * Assessment of comorbidities (Charlson score)
     * Screening for sarcopenia (using the SARC-F questionnaire),
     * An inventory of falls and their traumatic consequences,
     * Assessment of frailty status using FRIED criteria,
  2. Nutritional assessment :
     * nutritional status will also be asses
Other: Multicomponent exercise program — After inclusion in the protocol, participants with mobility disability risk factors are assigned to specialized and experienced kinesiologists at the end of the medical consultation.
  Patients will be invited to take part in group-based exercise sessions, in small groups of no more than 10 patients, under the supervision of a kinesiologist. There will be 20 sessions over 10 weeks, at a rate of 2 sessions per week, each lasting one hour. The Multicomponent exercise program included progressive resistance and balance training.
  Groups: Community-dwelling older adults assessed without mobility disability risk factors following initial
Other: Follow-up at T3 + 6 months and T3 + 12 months — Follow-up at T3 + 6 months :
  - After the T3 visit, patients will either be redirected to independent practice (booklet) or to relay structures. At T3 + 6 months (6 months after the 3-month visit), the kinesiologists will call each patient to assess their compliance with the program, any difficulties encountered, any falls (and their severity and consequences), fear of falling, their level of ADL/IADL autonomy, level of PA practice (RAPA), presence of frailty appreciation (FRIED), whether or not they have entered an institution.
  Follow-up at T3 + 12 months :
  At T3+12 months (12 months after the 3-month visit), patients will be seen again by the kinesiologists to make a final assessment of their physical and functional conditions, with measurements (Handgrip, SPPB, TUG, gait parameters, leg strength) and questionnaires (SarQol and FES-I).
  Patients will only be seen again by the kinesilogists, as this is mainly a check-up and final advice visit, to continue the exercises performed since.
  Groups: Community-dwelling older adults assessed without mobility disability risk factors following initial

SUMMARY:
The percentage of people aged over 80 will double in 25 years, reaching 10% of the population. This means that care practices for older adults will have to be adapted. Furthermore, disability-free life expectancy at 65 years old is 10.4 years, well below the overall life expectancy of 24.4 years for women and 19.1 years for men. Beneficiaries of the personalized autonomy allowance would increase by 60%, representing a major cost. Among the various factors predictive of loss of autonomy, loss of mobility and muscle weakness are major components (OR = 3.28 at 3 years) according to data from the latest meta-analyses. These two disability-causing factors are also responsible for multiple adverse events (falls, fractures, etc.), impaired quality of life and increased mortality. The only components accessible to preventive action and with a proven track record are exercise and nutrition. Despite a high level of evidence on the improvement of physical abilities and muscle strength, these programs are still not sufficiently implemented in practice. Indeed, neither the identification of seniors at risk of mobility disability, nor preventive actions are usually carried out in primary care. Setting up a care path, with personalized intervention combining, after identification, learning of good physical activity practices by a specialized kinesiologist and nutritional advice, followed by supervised exercise, for subjects at risk, is a public health imperative. The "Well on my legs" prevention program, supported by Hospices Civils de Lyon and present since 2014 in the Rhône region, is a concrete solution to this major public health challenge.

Analyses will be based on data collected through participant assessments during the "Well on my legs" prevention program. The analyses will make it possible to assess the risk factors of mobility disability in older adults at the start (T0) and at the end of the program (T3+12months), with the aim of improving the program's efficiency and evaluating its effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Patient covered by the "Well on my legs" program for primary and secondary prevention of mobility disability.

At least 1 of the following signs:

* Difficulty carrying a loaded shopping basket (load approx. 4.5 kg)
* Difficulty getting up from a chair without using arms
* Difficulty climbing a flight of stairs (10 steps)
* Difficulty moving around
* Slow gait speed
* Difficulty walking more than 400 meters without stopping
* Walking time < 30 min/d
* Fatigue during modest physical effort: shopping, housework,
* Fear of falling and/or at least one fall in the past year
* Recent involuntary weight loss: weight loss ≥ 5% in 1 month or BMI < 22kg/m2

Exclusion Criteria:

* - Patient who has not given consent to participate
* Patient under guardianship or legal protection in retrospective phase
* Patient with a locomotor handicap or SPPB <5
* Patient with a life expectancy of less than 12 months
* Patient with severe cognitive impairment
* Patient with exercise contraindications

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Community-dwelling older adults aged 70 and over, living at home, presenting risk factors for loss of mobility and having been assessed in the "Well on my legs" program for, at least, initial assessment (T0).
Sampling Method: Non-Probability Sample
Enrollment: 1600 (Estimated)
Dates: Start 2016-09-20 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
SPPB (Short Physical Performance Battery) | Change in the SPPB Score at 3 months of intervention and 1 year after
  Functional status is assessed by the overall Short Physical Performance Battery (SPPB) score, based on three components: gait speed, chair raising and balance tests.

CONTACTS AND LOCATIONS:
Overall Officials: DELAIRE Leo, Kinesiologist, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Service de médecine du vieillissement - Hôpital Edouard Herriot, Lyon, France, France